CLINICAL TRIAL: NCT02538627
Title: A Phase 1 Multi Arm Study Evaluating the Safety, Pharmacology and Preliminary Activity of the Co-Administration of MM-151 With Seribantumab (MM-121), Istiratumab (MM-141), or Trametinib in Biomarker-selected Cancer Patients
Brief Title: Phase 1 Combination Study of MM-151 With MM-121, MM-141, or Trametinib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-151-01-01-02
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: Heregulin-positive; EGFR; ErbB3; Phase I; Oncology; Cancer; IGF-1; MEKinhibitor; IGF-1R inhibitor; KRAS; NRAS
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — MM-151; seribantumab; Istiratumab; trametinib

ARMS (6):
- MM-151+MM-121 Dose Escalation (Experimental): MM-151 and MM-121 dose escalation in lung, head and neck, and colorectal cancers
  Interventions: Drug: MM-151; Drug: MM-121
- MM-151+ trametinib Dose Escalation (Experimental): MM-151 and trametinib dose escalation in lung, head and neck, and colorectal cancers.
  Interventions: Drug: MM-151; Drug: trametinib
- MM-151+MM-141 Dose Escalation (Experimental): MM-151 and MM-141 dose escalation in lung, head and neck, and colorectal cancers
  Interventions: Drug: MM-151; Drug: MM-141
- MM-151+trametinib Dose Escalation (Experimental): MM-151 and trametinib dose escalation in lung, head and neck, and colorectal cancers.
  Interventions: Drug: MM-151; Drug: trametinib
- Colorectal cancer Expansion (Experimental): Doses established in part 1 of the study
  Interventions: Drug: MM-151; Drug: MM-121; Drug: MM-141; Drug: trametinib
- Head and neck Expansion (Experimental): Doses established in part 1 of the study
  Interventions: Drug: MM-151; Drug: MM-121; Drug: MM-141; Drug: trametinib

INTERVENTIONS:
Drug: MM-151 — MM-151
Drug: MM-121 — MM-121
  Arms: Colorectal cancer Expansion; Head and neck Expansion; MM-151+MM-121 Dose Escalation
Drug: MM-141 — MM-141
  Arms: Colorectal cancer Expansion; Head and neck Expansion; MM-151+MM-141 Dose Escalation
Drug: trametinib — trametininb
  Other Names: MEKINIST
  Arms: Colorectal cancer Expansion; Head and neck Expansion; MM-151+ trametinib Dose Escalation; MM-151+trametinib Dose Escalation

SUMMARY:
This is a Phase 1 open-label, dose-escalation trial using "3+3" design, evaluating MM-151 co-administration with MM-121, MM-141, and trametinib at varying dose levels.

DETAILED DESCRIPTION:
This is a two-part Phase 1, non-randomized, open-label study of MM-151 plus MM-121, MM-141, or trametinib in patients with advanced, heregulin-positive lung, head and neck, and colorectal cancers. In part 1 of the study, cohorts of 3 or more patients will be treated at escalating doses of MM-151 in combination with MM-121, MM-141, and trametinib until a maximum tolerated combination dose for each combination is identified. In part 2 of the study, patients will be treated with the combination dose identified in part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >18 years of age
* Patients must be able to provide informed consent
* Willing to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of any study therapy). This applies to women of childbearing potential as well as fertile men and their partners
* Patients must be recovered from the effects of any prior surgery, radiotherapy or other antineoplastic therapy, up to CTCAE grade 1
* Patients must have either heregulin-positive cancer, cancer with RAS mutation, IGF-1 positive cancer, or RAS wild type cancer.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients who have an active infection or with an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, patients with tumor fever may be enrolled.)
* Patients with untreated (primary) or symptomatic CNS (primary or metastatic) malignancies; patients with CNS metastases who have undergone surgery or radiotherapy or who have been on a stable dose of corticosteroids for at least 2 weeks and whose disease is stable prior to the first scheduled day of dosing will be eligible for the trial.
* Patients who have received other recent antitumor therapy including any standard chemotherapy or radiation within 14 days (and having passed the time of any actual or anticipated toxicities) prior to the first scheduled dose of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
To find a phase II dose of MM-151 in combination with MM-121, MM-141, and trametinib based on maximum tolerated dose (MTD) in patients with lung, head and neck, and colorectal cancers | 1.5 years

SECONDARY OUTCOMES:
Number of dose limiting toxicities (DLTs) within a group | 1.5 years
Adverse event profile of MM-151 in combination with MM-121, MM-141, and trametinib | 1.5 years
Objective response to MM-151 in combination with MM-121, MM-141, and trametinib based on RECIST | 1.5 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado, Aurora, Colorado
  - Northside Hospital, Sandy Springs, Georgia
  - Northwestern, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Vanderbilt, Nashville, Tennessee